CLINICAL TRIAL: NCT07347262
Title: A Pilot Study Evaluating the Use of a Novel Noninvasive Breath Test to Identify Patients at Risk for Developing Gestational Diabetes
Brief Title: A Study Using Breath Tests to Identify Patients at Risk for Gestational Diabetes
Status: Completed | Type: Observational
Sponsor: Kaplan Medical Center (Other)
Collaborators: University of Galway (Other)
Responsible Party: Principal Investigator, Maya Oberman, Attending physician, Kaplan Medical Center
Other Study IDs: 0116-19-KMC
Record Dates: First submitted 2023-09-21; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Noninvasive Breath Test in Order to Identify Patients at Risk for Developing Gestational Diabetes — After a short explanation on how to use the kit participants will be asked to sample their breath every 15 minutes starting 30 minutes before the ingestion of glucose and ending six hours after the ingestion.

SUMMARY:
The aim of our study is to evaluate the feasibility, and diagnostic value of oral 13C labelled glucose breath test compared to the GCT and OGTT tests.

DETAILED DESCRIPTION:
This prospective observational pilot study will include pregnant patients with a singleton fetus up to 33 weeks gestation.

Patients meeting the inclusion criteria who are willing to participate will be asked to drink 50 or 100 grams of glucose in 200 ml water (disposable plastic cup). The test will start at approximately 08:00 with no change in normal diet is needed prior to the GCT, or after an 8-14 hour overnight fast for the OGTT.

The test will be performed at the Maternal Fetal Medicine outpatient clinics, the Maternal Fetal Medicine unit for inpatients or at the patient's residence.

Samples collection

Glucose samples:

1. Venous blood samples to measure serum glucose levels will be drawn at a timing according to the performed test: for GCT at one hour after the ingestion of glucose (standard 50 grams GCT) and for OGTT at to, t1, t2 and t3 (standard 100 grams OGTT).
2. Finger prick glucometer (DEX) readings will be done at one and two hours after the ingestion of glucose for participants completing GCT.

Each participant will receive a kit containing 30 12ml exetainers (Labco, UK), a compatible strew and a stamped envelope (addressed to OBGYN department, Kaplan Medical Center, Rehovot). The exetainers will be numbered sequentially and marked by the participant code (initials and participant number). After a short explanation on how to use the kit participants will be asked to sample their breath every 15 minutes starting 30 minutes before the ingestion of glucose and ending six hours after the ingestion. Patients who are taking the test at the Maternal Fetal Medicine clinic will be asked to remain at the clinic for the duration of six hours, until completing all of the samples. Patients who are taking the test while admitted to the Maternal Fetal Medicine ward and are due for discharge will not be delayed as discharge is usually until 14:00. During the six hours of participation patients will be ask to avoid food or drink. Afterwards, participants will keep the envelope in their home until a pickup is coordinated by a member of the research team.

Samples can be kept up to three months before being processed. The coded samples will next be sent to Amir Shafat's lab at Ireland for processing. Samples will be analyzed on a continuous-flow Isotope Ratio Mass Spectrometer (ABCA, Serco, UK) for breath CO2 enrichment against Vienna-Pee Dee Belemnite, a known international standard for 13C. Enrichment will be expressed in atom fraction and δV-PDB. Pilot data in Amir's lab demonstrated that this procedure gives excellent resolution of breath enrichment (to within 1 part per million) and includes peak excretion of 13CO2 in all volunteers. Percent dose recovered and other parameters indicating the rate of glucose oxidation will be calculated from the enrichment curve. Amir's laboratory has extensive experience in stable isotope and breath testing.

A few days (and no longer than one week) after the test participants will receive their GCT or OGTT result by phone and fax/email. Participants will be asked to present the test result to their physician in the next prenatal visit. For participants with a pathological GCT score, >139 mg/dL, a letter will be sent to the attending physician requesting to perform the 100 grams OGTT either as part of the study or at the health care provider clinic. Participants with one or more elevated glucose values in the OGTT, will be asked to contact their physician as soon as possible for further guidance. Two weeks after the test, a follow-up phone call will be done to all participants with a pathological result in order to ensure that the OGTT had been completed and to record the OGTT result in case of a pathological GCT, or to ensure the appropriate surveillance has begun in case of a pathological OGTT.

Demographic data including: a) maternal age; b) maternal height: c) pre-pregnancy and current weight; d) obstetrical history e) background medical illnesses and medications.

Sample size estimation In this pilot study the investigators aim to recruit 50 participants in each group (GCT and OGTT) out of which it is expected that 8-11 will have pathological result (16-21% pathological GCT).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* ages 18 to 45 years old
* A singleton pregnancy
* Confirmed gestational age by a documented first-trimester ultrasound.

Exclusion Criteria:

* Patients below the age of 18 or above 45 years-old
* Patients diagnosed with gestational or pre-gestational diabetes
* Patients with multiple pregnancies or fetuses with congenital and/or chromosomal anomalies
* Patients after a multifetal pregnancy reduction (spontaneous or iatrogenic)
* Patients not having a sonographic dating during the first trimester of pregnancy
* Patients with conditions or medications that affect glucose metabolism
* Patients who will refuse to consent, or are not fit or able to read, understand, or sign an informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This prospective observational pilot study will include pregnant patients with a singleton fetus up to 33 weeks gestation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
The aim of our study is to evaluate the feasibility of oral 13C labelled glucose breath test compared to the GCT and OGTT tests. | At the time of the glucose tolerance test (GCT/ OGTT)
  We will assess feasibility via recruitment and test completion.
To evaluate the diagnostic value of oral 13C labelled glucose breath test compared to the GCT and OGTT tests. | At the time of the glucose tolerance test (GCT/ OGTT)
  We will assess agreement between exogenous glucose oxidation (breath test) and blood glucose (OGTT).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Background] O'Sullivan JB, Mahan CM, Charles D, Dandrow RV. Screening criteria for high-risk gestational diabetic patients. Am J Obstet Gynecol. 1973 Aug 1;116(7):895-900. doi: 10.1016/s0002-9378(16)33833-9. No abstract available. PMID 4718216
- [Background] Carpenter MW, Coustan DR. Criteria for screening tests for gestational diabetes. Am J Obstet Gynecol. 1982 Dec 1;144(7):768-73. doi: 10.1016/0002-9378(82)90349-0. PMID 7148898
- [Background] Roeckner JT, Sanchez-Ramos L, Jijon-Knupp R, Kaunitz AM. Single abnormal value on 3-hour oral glucose tolerance test during pregnancy is associated with adverse maternal and neonatal outcomes: a systematic review and metaanalysis. Am J Obstet Gynecol. 2016 Sep;215(3):287-97. doi: 10.1016/j.ajog.2016.04.040. Epub 2016 Apr 29. PMID 27133007
- [Background] van Leeuwen M, Louwerse MD, Opmeer BC, Limpens J, Serlie MJ, Reitsma JB, Mol BW. Glucose challenge test for detecting gestational diabetes mellitus: a systematic review. BJOG. 2012 Mar;119(4):393-401. doi: 10.1111/j.1471-0528.2011.03254.x. Epub 2012 Jan 20. PMID 22260369
- [Background] Goldberg RJ, Ye C, Sermer M, Connelly PW, Hanley AJ, Zinman B, Retnakaran R. Predictors and clinical implications of a false negative glucose challenge test in pregnancy. J Obstet Gynaecol Can. 2013 Oct;35(10):889-898. doi: 10.1016/S1701-2163(15)30810-0. PMID 24165056
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Harlass FE, Brady K, Read JA. Reproducibility of the oral glucose tolerance test in pregnancy. Am J Obstet Gynecol. 1991 Feb;164(2):564-8. doi: 10.1016/s0002-9378(11)80021-9. PMID 1992702
- [Background] Heise T, Zijlstra E, Nosek L, Heckermann S, Plum-Morschel L, Forst T. Euglycaemic glucose clamp: what it can and cannot do, and how to do it. Diabetes Obes Metab. 2016 Oct;18(10):962-72. doi: 10.1111/dom.12703. Epub 2016 Jul 13. PMID 27324560
- [Background] Huhn EA, Rossi SW, Hoesli I, Gobl CS. Controversies in Screening and Diagnostic Criteria for Gestational Diabetes in Early and Late Pregnancy. Front Endocrinol (Lausanne). 2018 Nov 27;9:696. doi: 10.3389/fendo.2018.00696. eCollection 2018. PMID 30538674
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes. Diabetes Care. 2017 Jan;40(Suppl 1):S11-S24. doi: 10.2337/dc17-S005. No abstract available. PMID 27979889
- [Background] Dillon EL, Janghorbani M, Angel JA, Casperson SL, Grady JJ, Urban RJ, Volpi E, Sheffield-Moore M. Novel noninvasive breath test method for screening individuals at risk for diabetes. Diabetes Care. 2009 Mar;32(3):430-5. doi: 10.2337/dc08-1578. Epub 2008 Dec 15. PMID 19074994
- [Background] Schellekens RC, Stellaard F, Woerdenbag HJ, Frijlink HW, Kosterink JG. Applications of stable isotopes in clinical pharmacology. Br J Clin Pharmacol. 2011 Dec;72(6):879-97. doi: 10.1111/j.1365-2125.2011.04071.x. PMID 21801197
- [Background] Koletzko B, Sauerwald T, Demmelmair H. Safety of stable isotope use. Eur J Pediatr. 1997 Aug;156 Suppl 1:S12-7. doi: 10.1007/pl00014267. PMID 9266209
- [Background] Gregg CT. Some application of stable isotopes in clinical pharmacology. Eur J Clin Pharmacol. 1974 Jul 26;7(4):315-9. doi: 10.1007/BF00560350. No abstract available. PMID 4605121
- [Background] Hsu HW, Butte NF, Wong WW, Moon JK, Ellis KJ, Klein PD, Moise KJ. Oxidative metabolism in insulin-treated gestational diabetes mellitus. Am J Physiol. 1997 Jun;272(6 Pt 1):E1099-107. doi: 10.1152/ajpendo.1997.272.6.E1099. PMID 9227457
- [Background] Ranawana V, Clegg ME, Shafat A, Henry CJ. Postmastication digestion factors influence glycemic variability in humans. Nutr Res. 2011 Jun;31(6):452-9. doi: 10.1016/j.nutres.2011.05.006. Epub 2011 Jun 17. PMID 21745627
- [Background] Morey S, Shafat A, Clegg ME. Oral versus intubated feeding and the effect on glycaemic and insulinaemic responses, gastric emptying and satiety. Appetite. 2016 Jan 1;96:598-603. doi: 10.1016/j.appet.2015.11.002. Epub 2015 Nov 10. PMID 26551790
- [Background] Thondre PS, Shafat A, Clegg ME. Molecular weight of barley beta-glucan influences energy expenditure, gastric emptying and glycaemic response in human subjects. Br J Nutr. 2013 Dec;110(12):2173-9. doi: 10.1017/S0007114513001682. Epub 2013 Jun 7. PMID 23742725
- [Background] Clegg ME, Shafat A. The effect of agar jelly on energy expenditure, appetite, gastric emptying and glycaemic response. Eur J Nutr. 2014;53(2):533-9. doi: 10.1007/s00394-013-0559-x. Epub 2013 Jul 20. PMID 23872837
- [Background] Sevket O, Ates S, Uysal O, Molla T, Dansuk R, Kelekci S. To evaluate the prevalence and clinical outcomes using a one-step method versus a two-step method to screen gestational diabetes mellitus. J Matern Fetal Neonatal Med. 2014 Jan;27(1):36-41. doi: 10.3109/14767058.2013.799656. Epub 2013 May 30. PMID 23617557
- [Background] Olagbuji BN, Aderoba AK, Kayode OO, Awe CO, Akintan AL, Olagbuji YW; Gestational Diabetes Study Group-Nigeria. Accuracy of 50-g glucose challenge test to detect International Association of Diabetes and Pregnancy Study Groups criteria-defined hyperglycemia. Int J Gynaecol Obstet. 2017 Dec;139(3):312-317. doi: 10.1002/ijgo.12304. Epub 2017 Sep 14. PMID 28833075
- [Background] Arbib N, Gabbay-Benziv R, Aviram A, Sneh-Arbib O, Wiznitzer A, Hod M, Chen R, Hadar E. Third trimester abnormal oral glucose tolerance test and adverse perinatal outcome. J Matern Fetal Neonatal Med. 2017 Apr;30(8):917-921. doi: 10.1080/14767058.2016.1190825. Epub 2016 Jun 8. PMID 27186963